CLINICAL TRIAL: NCT07246005
Title: A Randomised Pilot Study Assessing the Optimal Duration of Anticoagulation for Left Ventricular Thrombus
Brief Title: LVT DURATION: Pilot Study of Anticoagulation Duration for Left Ventricular Thrombus
Acronym: LVT Duration
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1008221; G-002409 (Other Grant/Funding Number: Barts Charity)
Record Dates: First submitted 2025-10-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Left Ventricular Thrombus
Keywords: LVT; Left Ventricular Thrombus; Thrombus; Thrombi; anticoagulant
MeSH Terms: conditions — Thrombosis | interventions — apixaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continue pre prescribed rivaroxaban or apixaban or warfarin (Experimental): If randomised to this arm, participants will continue on their rivaroxaban or apixaban or warfarin for the study related time period.
  Interventions: Drug: Continue rivaroxaban or apixaban or warfarin
- Discontinue pre prescribed rivaroxaban or apixaban or warfarin (Experimental): If randomised to this arm, patients (who have already been on OAC for a period of 3 months) will discontinue their rivaroxaban or apixaban or warfarin.
  Interventions: Drug: Discontinue rivaroxaban or apixaban or warfarin

INTERVENTIONS:
Drug: Continue rivaroxaban or apixaban or warfarin — The study is asessing the impact of discontinuation of oral anticoagulation in patients with LV thrombus diagnosis.
  Arms: Continue pre prescribed rivaroxaban or apixaban or warfarin
Drug: Discontinue rivaroxaban or apixaban or warfarin — discontinue rivaroxaban or apixaban or warfarin
  Arms: Discontinue pre prescribed rivaroxaban or apixaban or warfarin

SUMMARY:
The LVT DURATION (Optimal Duration of Anticoagulation for LV Thrombus) is a pilot study planned to assess the practicalities of conducting a randomised control trial (RCT) whilst establishing data around the ideal duration of anticoagulation in the treatment of LV thrombus. The main objectives of the study are:

* To assess the practicalities of conducting an RCT with regard to recruitment, retention, and outcome measurement.
* To identify the optimal length of anticoagulation in the treatment of LV Thrombus

After randomisation participants will:

* Continue their prescribed oral anticoagulant for the remainder of the trial
* Discontinue their prescribed oral anticoagulant for the remainder of the trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LV thrombus less than 12 months ago
* On Apixaban at the time of randomisation
* Completed at least 3 months of anticoagulation treatment for LV thrombus
* Persistent laminar/ mural thrombus or persistent LV dysfunction

Exclusion Criteria:

* Any clinical condition requiring long term anticoagulation treatment as per investigator's judgement.
* SSE since LV thrombus diagnosis
* Contraindication to continuing anticoagulation therapy
* Non-ischaemic Cardiomyopathy
* Age less than 18 years
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Stroke and Systemic Embolism (SSE) | 6 months
  Number of SSE events following randomisation
All-Cause Mortality | 6 months
  Number of deaths from any cause following randomisation

SECONDARY OUTCOMES:
Major Bleeding | 6 months
  Rates of major bleeding (BARC ≥ 3) events following randomisation.
Minor Bleeding | 6 months.
  Rates of minor bleeding (BARC ≤ 2) events following randomisation.
New LV Thrombi | 6 months
  Rates of new LV thrombus formation between the groups.
Resolved Thrombus | 6 months
  Rates of LV thrombus resolution between the groups.
Hospitalisation | 6 months
  Total number of days in hospital between continuing versus stopping anticoagulation.
Cost Comparison | 6 months
  Total measured costs between continuing versus stopping anticoagulation.
MI | 6 months
  Number of participants experiencing MI following randomisation
EQ-5D-5L | 6 months
  Quality of life of participants measured by EQ-5D-5L.
Perspectives of Clinicians and Patients | 6 months
  Qualitative assessment of clinician and patient views on study design, procedures, and relevance, collected via structured interviews and surveys
Target Vessel Revascularization (TVR) | 6 months
  Number of participants undergoing TVR following randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided